CLINICAL TRIAL: NCT03289598
Title: A Cluster Randomised Feasibility Trial Evaluating Involving Community-dwelling Older Adults in Activities in Relation to Meals in a Rehabilitation Program; Recruitment, Data Collection and Protocol
Brief Title: Effect of Involving Community-dwelling Older Adults in Activities in Relation to Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Danish Dietetic Association (Other)
Collaborators: The Danish Meal Partnership (Unknown); Ministry of Environment and Food of Denmark (Unknown); Metropolitan University College (Other); National Board of Health, Denmark (Other Government); The City of Odense (Unknown); Danish Diet & Nutrition Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PROJECT_APM
Record Dates: First submitted 2017-09-16; First posted 2017-09-21 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2018-08

CONDITIONS: Frail Older Adults
MeSH Terms: interventions — Meals

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventionsgroup (Experimental)
  Interventions: Behavioral: A rehabilitation process involving collaborative goal setting with a case manager about managing own food and meals
- Controlgroup (No Intervention)

INTERVENTIONS:
Behavioral: A rehabilitation process involving collaborative goal setting with a case manager about managing own food and meals — The intervention consists of two parts:
  1. Education of the health care staff with three day's education focusing of aspects of food, meals and nutrition to old people.
  2. The individual participants in the intervention group will be participating in a rehabilitation process involving collaborative goal setting with a case manager. All the case managers have a background as registered dietician and will before start of the intervention be trained in managing a rehabilitation process with focus on meals and food. The training will consist of three days of education in, respectively, areas in relation to rehabilitation and the role as a care manager. Specific topics include; assessment of functional abilities in relation to meals and food; goal setting by means of GAS (Goal Attainment Scaling), ethical considerations and communication.
  Arms: Interventionsgroup

SUMMARY:
Community-dwelling older adults receiving support at home such as meals-on-wheels may lose the ability to preserve social, cognitive, and functional abilities, when becoming accustomed to and dependent of community aged care. When still able to cook older adults often hold some control over the foods that are prepared and which they eat, and which helps to foster identity. The purpose of this study is to evaluate community-dwelling older adults being involved in activities in relation to meals in a rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling older people (64+ years)
* Able to eat and drink
* Receive meals-on-wheels from the municipality at the time of recruitment
* Live in the city of Odense

Exclusion Criteria:

* Moderate-severe dementia as judged by the home -care staff
* Being deaf and/or not understand the language of Danish.
* Not being able to sign the informed consent
* Receiving (or likely to receive in the next 6 months) enteral tube feeding or parenteral nutrition;
* Participating in other project in the municipality about nutritional support in the form of dietetic advice;
* Or on an end-of-life care pathway

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Quality of life | Up to 6 months
  EuroQol (EQ-5D) is a questionnaire with five questions to be answered in three categories of movement, self-care, usual activities, pain/discomfort and anxiety/depression.

SECONDARY OUTCOMES:
30 seconds chair-stand | Up to 6 months
  30 seconds chair-stand will be used to measure muscle strength. Participants are asked to fold their arms across their chest and to stand up and sit down on a chair without pushing off with arms, as many times as possible for 30 seconds.
Weight | Up to 6 months
  Weight in kilograms
Height | Up to 6 months
  Height in meter and centimetre
Loneliness | Up to 6 months
  Loneliness will be measured by the UCLA Loneliness Scale. The scale consists of 20 items (11 positive and 9 negative), describing subjective feelings of loneliness.
Mental well-being | Up to 6 months
  Mental well-being will be measured by the short Warwich-Edinburgh Mental Well-being Scale (SWEMWBS) - Danish version 2014. SWEMWBS is a 7-item scale; each answered on a 1 to 5 Likert scale, with most items representing aspects of psychological and eudemonic well-being, and few covering hedonic well-being or affect.
Self-efficacy | Up to 6 months
  Self-efficacy will be measured by The General Self-Efficacy Scale (GSE).The GSE is a 10-item psychometric scale will be used to assess optimistic self-beliefs to cope with a variety of difficult demands in life.
Satisfaction with food-related life | Up to 6 months
  The satisfaction with food-related life will be measured by the Satisfaction with Food-related Life (SWFL) scale.The SWFL, consists of 5 items grouped into a single dimension (e.g. Food 1: Food and meals are positive elements; Food 2: I am generally pleased with my food; Food 3: My life in relation to food and meals is close to ideal; Food 4: With regards to food, the conditions of my life are excellent; Food 5: Food and meals give me satisfaction in daily life.). In each scale, the respondents must indicate their degree of agreement with these statements using a 6-level Likert scale (1 = disagree completely, 6 = agree completely).

CONTACTS AND LOCATIONS:
Overall Officials: Mette Pedersen, Study Director — The Danish Dietetic Association
Locations (1):
- The Danish Dietetic Association, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Husted MM, Beck AM, Ulrikkeholm LK. A cluster randomised feasibility pilot trial evaluating involving community-dwelling older adults in activities in relation to meals in a rehabilitation program; recruitment, data collection and protocol. Pilot Feasibility Stud. 2018 Aug 6;4:134. doi: 10.1186/s40814-018-0323-3. eCollection 2018. PMID 30123525